CLINICAL TRIAL: NCT02092974
Title: Mechanism of tDCS-induced Learning Enhancement - the Role of Serotonin
Acronym: LESO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LESO
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Healthy Young and Older Adults
Keywords: transcranial direct current stimulation (tDCS); selective serotonin reuptake inhibitor (SSRI); young; older adults
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- tDCS + SSRI (Experimental)
  Interventions: Procedure: tDCS; Drug: Citalopram
- tDCS + placebo (Placebo Comparator)
  Interventions: Procedure: tDCS
- sham-tDCS + SSRI (Sham Comparator)
  Interventions: Drug: Citalopram
- sham-DCS + placebo (Placebo Comparator)
  Interventions: Other: sham-tDCS + placebo

INTERVENTIONS:
Procedure: tDCS
  Other Names: transcranial direct current stimulation
  Arms: tDCS + SSRI; tDCS + placebo
Drug: Citalopram
  Other Names: SSRI
  Arms: sham-tDCS + SSRI; tDCS + SSRI
Other: sham-tDCS + placebo
  Arms: sham-DCS + placebo

SUMMARY:
The aim of this study is to assess whether the application of a selective serotonin reuptake inhibitor (SSRI) enhances and prolongs the learning enhancement achieved by anodal transcranial direct current stimulation (atDCS). For this, young and older healthy subjects will be tested with a well established learning paradigm. Results of this study may help to support the application of atDCS also in patients, e.g. with dementia or mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* right handedness
* unobtrusive neuropsychological screening
* ability to provide written informed consent
* no pathological findings in head MRI
* age: 18 to 35 years (young adults) or 50-80 years (older adults)
* Highly effective contraception (Pearl Index < 1) or reliable abstinence from any heterosexual relationships in women of childbearing potential

Exclusion Criteria:

* severe internal or psychiatric disease (especially depression or suicidal thoughts)
* epilepsy
* cognitive impairment (< SD under age adjusted norm in neuropsychological testing)
* concurrent taking of serotonin precursors (tryptophan, 5-HTP) or MAO inhibitors
* concurrent taking of tramadol or triptans
* concurrent taking of pimozide or linezolid
* concurrent taking of other drugs prolonging the QT-interval
* long-QT-syndrome
* hypokalemia or hypomagnesemia
* known intolerance of the study medication
* claustrophobia or metallic implants, tattoos (MRI exclusion criteria)
* pregnancy or lactation
* participation in another drug-interventional clinical trial within the last month or during the entire study
* probands that are placed in an institution due to official or judicial order
* non-agreement to save and transmit pseudonymised study data within the clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Recall score after learning under tDC stimulation + SSRI compared to learning under tDC stimulation + placebo. | immediately after end of learning phase (approx. 1 hour)
  Recall score immediately after learning phase (=training of visual-spatial abilities) under tDC stimulation + SSRI application compared to learning under tDC stimulation + placebo.

SECONDARY OUTCOMES:
prolongation of the atDCS induced learning enhancement by SSRI | 1 week
  Measurement of recall scores on the evening of the same day after the learning phase (+tDCS + SSRI), the morning of the day after and 1 week later in order to assess the prolongation of atDCS induced learning enhancement by the SSRI.
Increase of learning enhancement by atDCS + placebo or sham-tDCS + SSRI vs. sham-tDCS + placebo | immediately after learning phase (approx. 1 hour)
  Measurement of recall scores directly after learning phase after application of atDCS + placebo or sham-tDCS + SSRI vs. sham-tDCS + placebo.
prolongation of learning enhancement by atDCS + placebo or sham-tDCS + SSRI vs. sham-tDCS + placebo | 1 week
  Measurement of recall scores on the evening of the same day of learning phase, the morning of the day after and 1 week later under application of atDCS + placebo or sham-tDCS + SSRI vs. sham-tDCS + placebo, in order to assess prolongation of learning enhancement by SSRI.
genotyping of learning related polymorphisms | once
  To assess predictors of SSRI-enhanced brain stimulation, genotyping of several learning related polymorphisms will be performed (i.e., APOE, BDNF, Val66Met, COMT, Val158Met, KIBRA, rs17070145, 5-Hydroxytryptamine transporter).

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Result] Prehn K, Stengl H, Grittner U, Kosiolek R, Olschlager A, Weidemann A, Floel A. Effects of Anodal Transcranial Direct Current Stimulation and Serotonergic Enhancement on Memory Performance in Young and Older Adults. Neuropsychopharmacology. 2017 Jan;42(2):551-561. doi: 10.1038/npp.2016.170. Epub 2016 Aug 24. PMID 27555381